CLINICAL TRIAL: NCT06094959
Title: Integrating Suicide Prevention Packages Into Task-shifted Mental Health Interventions in Low-resourced Contexts
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: Dhulikhel Hospital, Kathmandu University School of Medical Sciences (Unknown); American Foundation for Suicide Prevention (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 2000029480; No NIH funding (Other: 9.20.23 CB)
Record Dates: First submitted 2023-10-13; First posted 2023-10-23 (Actual); Last update posted 2024-10-29 (Actual); Status verified 2024-10

CONDITIONS: Suicide Prevention
MeSH Terms: conditions — Suicide Prevention

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Suicide Prevention Package — The implementation package consists of co-designed and culturally adapted suicide prevention elements including suicide crisis response planning, contact follow up phone calls, and healthcare provider support mechanisms to optimize implementation.

SUMMARY:
The goal of this study is to assess the feasibility and acceptability of implementing a co-designed suicide prevention package of implementation strategies (SuPP) in a pilot open, non-randomized, clinical trial. The main questions it aims to answer are:

1. What is the feasibility of implementing the SuPP open clinical trial?
2. What is the degree to which SuPP was implemented correctly
3. What is the perceived acceptability of SuPP among providers and patients?

Participants will include healthcare providers and patients at risk for suicide. Providers will identify and provide culturally adapted safety planning and contact follow up to at-risk patients over a period of six months. Patients will receive an initial culturally adapted patient-centered safety plan and receive a tapered series of contacts (phone calls) over the course of six months from health providers.

DETAILED DESCRIPTION:
Low and middle income countries (LMIC) hold 75% of the world's suicides. Suicide disproportionately affects those living in poverty and in adverse conditions and, in LMIC settings, up to 20% of maternal deaths are due to suicide. In Nepal, suicide is a leading cause of death among women of reproductive age. Despite the disproportionate burden, systematic suicide detection and prevention mechanisms are nearly non-existent. Deaths are only a fraction of the burden, where evidence from Nepal reports between 5 and 27% of individuals have current thoughts of suicide. Suicidal behavior remains under-reported and is difficult for clinicians to properly identify and monitor, especially in limited health systems. This calls for improved understanding of how to identify and monitor individuals at risk for suicidal behavior. Therefore, this study seeks to integrate existing hospital healthcare providers into suicide prevention, contributing much needed evidence for multi-pronged, accessible strategies to reduce a leading cause of death worldwide.

This study's purpose is to adapt and pilot the implementation of packaged suicide prevention strategies in a low-resource setting. The impact involves informing an implementation plan to test in a fully powered future trial. Findings will contribute to the evidence of systems-integrated suicide prevention strategies and result in a multi-level package for mental health service integration that can be utilized around the world. Ultimately, this project will save lives and improve under-resourced health systems. The pilot trial is not powered for statistical analysis, but data will be monitored monthly and continuously analyzed to facilitate iterative revision, then finalization of the protocol.

The implementation package to be tested (the Suicide Prevention Package, SuPP) will include a culturally adapted suicide crisis response plan and a series of contacts via phone call from a hospital healthcare provider. This is a small open, non-randomized, pilot trial to assess the feasibility and acceptability of SuPP within the existing health system. The investigators will select delivery agents, an implementation strategy, and complete SuPP training. The investigators will train the selected delivery agents and their supervisory team (e.g., hospital nurses, physicians, and department heads) in SuPP (detection, safety planning, brief contact follow up). Participants will be recruited through the hospital's emergency department. Following suicide risk detection (e.g., suicide attempt in the past 6 months), 24 at-risk patients will be enrolled in the open trial and given the full SuPP package. All participants will receive standard of care, the SuPP package is in addition. In accordance with recommendations for pilot trial studies, The investigators have established qualitative and quantitative indicators to guide decisions about what procedures to carry through to the full trial and when modifications should be made. Each patient will be provided contact and suicide crisis response planning (weekly, then tapering to monthly) for at least 6 months. SuPP feasibility and acceptability will be determined by the following criteria: delivery agent fidelity to SuPP elements at 75% or greater; retention of at least 70% of participants through 6 months of SuPP; fewer than 15% missing items on outcome measures across all assessments; 80% of delivery agents and patients finding SuPP acceptable. In domains where criteria are met, the investigators will retain the procedure for a future full trial. In domains where criteria are not met, the investigators will modify procedures for the future full trial.

ELIGIBILITY:
Inclusion Criteria (healthcare workers):

* Be older than 18 at the time of recruitment
* Speak Nepali fluently
* Be actively employed by Dhulikhel Hospital/KUSMS
* Have a valid certificate of practice from the Ministry of Health and Population

Exclusion Criteria (healthcare workers)

* Have less than 3 months of experience in current position
* Be planning to remain in the study area or current position for less than six months
* Be unable to provide voluntary informed consent for any reason

Inclusion Criteria (trial patients):

* Speak Nepali fluently
* Be older than 18 at the time of recruitment
* Be actively receiving care from a KUDH clinician
* Permanently reside in Dhulikhel District
* Have access to a cell phone
* Screen positive for suicide risk

Exclusion Criteria (trial patients):

* Reside outside of the catchment area
* Be planning to leave relocate their residence in the next 6 months
* Unable to provide voluntary informed consent for any reason
* Unable to provide a mobile phone number for contact
* Present evidence of active and untreated mania or psychosis that could interfere with the participant's ability to volitionally consent to research or interfere with their ability to safely and reliably complete research

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2023-05-30 (Actual); Primary Completion 2024-07-08 (Actual); Study Completion 2024-07-23 (Actual)

PRIMARY OUTCOMES:
Feasibility assessed by recruitment | 6 months post intervention
  Recruitment defined as the percent of eligible participants that agree to participate
Feasibility assessed by treatment adherence | 6 months post intervention
  The percent of participants that completed one session with the intervention delivery agent
Feasibility assessed by treatment adherence- SuPP | 6 months post intervention
  Treatment adherence defined as the percent of participants who remain in SuPP
Feasibility assessed by retention | 6 months post intervention
  The percent of participants who completed all follow up measures
Feasibility assessed by retention- missing items | 6 months post intervention
  The percent of missing measure items per participant
Feasibility assessed by screening | 6 months post intervention
  The number of participants screened and referred
Percent enrolled | 6 months post intervention
  The percent of referred participants that enrolled
Median number of sessions completed | 6 months post intervention
  Median number of sessions completed

SECONDARY OUTCOMES:
Acceptability assessed by Consolidated Framework for Implementation Research (CFIR) qualitative interviews | 6 months post intervention
  CFIR interviews are qualitative interviews that will be thematically analyzed with qualitative analysis guided by the CFIR framework and taxonomy.

CONTACTS AND LOCATIONS:
Overall Officials: Ashley Hagaman, PhD, Principal Investigator — Yale University
Locations (1):
- Dhulikhel Hospital, Dhulikhel, Nepal

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Shrestha AP, Shrestha R, Risal A, Shakya R, Sigdel K, Bajracharya R, Paudel P, Gumudavelly D, Egger E, Zhuang S, Vijayakumar L, Hagaman A. Evaluating implementation preparedness for suicide screening and referral in a Nepali emergency department: A mixed-methods study. Implement Res Pract. 2025 Jul 6;6:26334895251343644. doi: 10.1177/26334895251343644. eCollection 2025 Jan-Dec. PMID 40630920